CLINICAL TRIAL: NCT01430130
Title: Investigation of a Novel Mechanomodulating Polymer to Maximize the Outcomes of Scar Revision Procedures
Brief Title: Investigation of a Novel Silicone Dressing to Maximize the Outcomes of Scar Revision Procedures (IMPROVE)
Acronym: IMPROVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neodyne Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CA005
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Results first posted 2014-11-28 (Estimated); Last update posted 2014-11-28 (Estimated); Status verified 2014-11

CONDITIONS: Hypertrophic
Keywords: scar; incision; wound healing; scarring; scar revision
MeSH Terms: conditions — Hypertrophy; Cicatrix; Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All Study Participants (Experimental): Half of the revised incision was treated with the embrace device. Half of the revised incision was treated according to the Investigator's standard of care. Participant served as his/her own control.
  Interventions: Device: embrace device

INTERVENTIONS:
Device: embrace device — Adhesive bandage/dressing intended to minimize scar formation.
  Other Names: Neodyne dressing

SUMMARY:
Neodyne has developed an investigational dressing for post-operative incision care. Neodyne is conducting this research to study whether the investigational dressing, called the Neodyne Dressing, can minimize scar formation in a simple manner.

DETAILED DESCRIPTION:
It is proposed to study a dressing designed to reduce the appearance of scars after scar revision surgery. It is expected that by managing the incision site after primary closure but during the longer term healing phase, scar formation may be minimized.

ELIGIBILITY:
Inclusion Criteria:

* The scar to be revised is:

  * at least 12 months old
  * linear and suitable for revision by excision and direct closure
  * appropriate size and location for Neodyne Dressing
* The subject:

  * age > 18 and < 65 years old

Exclusion Criteria:

* Subjects with a skin disorder that is chronic or currently active.
* Subjects who are involved in ongoing litigation in connection with the scar to be revised.
* Subjects with a history of collagen vascular disease
* Subjects diagnosed with scleroderma
* Subject who currently smokes
* Subjects with known adverse reactions to steri-strip tapes, medical tapes, or adhesives
* Subjects with oozing, dehiscence, non-closed/healed incisions at time of first application.
* Subjects with inability to maintain adequate care of incision.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Weintraub, MD, Principal Investigator — Duet Plastic Surgery; Angeline Lim, MD, Principal Investigator — Duet Plastic Surgery
Locations (1):
- Duet Plastic Surgery, Palo Alto, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All procedures were performed at a single outpatient surgery clinic between September of 2011 and May of 2012.
Period: Overall Study
Arm/Group | All Study Participants
Started | 12
Completed | 10
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Infection on Control Side of Incision | 1

BASELINE CHARACTERISTICS:
Population: After meeting all eligibility criteria, 12 patients were enrolled.
Arm/Group | All Study Participants
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogue Scale (VAS)
Description: Visual Analogue Scale Scar Score (VAS Scar Score) was defined and validated by Duncan et al 2006[1]. This scale consists of a 10cm line representing scar quality, with 0 representing normal skin and 10 indicating a poor scar. The assessor places a mark along the line to represent the appearance of the scar. This mark is translated into a score by measuring its position on the 10cm line to one decimal place. The independent panel used this to scale the primary outcome.
  [1] Duncan J, Bond J, Mason T, Ludlow A, Cridland P, O'Kane S and Ferguson M. Visual Analogue Scale Scoring and Ranking: A Suitable and Sensitive Method for Assessing Scar Quality? Plast. Reconstr. Surg. 118: 909, 2006.
Time Frame: 6 months
Population: Per protocol, all eligible patients who did not exit the study prematurely.
Measure: Mean (Standard Error); unit: Units on a scale
Groups:
- Treated Side: Half of the revised incision was treated with the embrace device.
- Control Side: Half of the revised incision was treated according to the investigator's standard of care. Participant served as his own control.
Arm/Group | Treated Side | Control Side
Number analyzed (Participants) | 10 | 10
Units on a scale | 3.78 (0.35) | 5.58 (0.39)

2. Secondary Outcome: Subject and Investigator Satisfaction With the Aesthetic Results
Time Frame: Up to 12 months
Reporting Status: Not Posted

3. Secondary Outcome: Ease of Use
Time Frame: Up to 12 months
Reporting Status: Not Posted

4. Secondary Outcome: Comfort Level Related to Study Device Application, Wear and Removal
Time Frame: Up to 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Comparison of Scar Smoothness of Treated Side as Compared to the Control Side
Time Frame: Up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse Events were reported via phone call or in person at weekly site visits for Neodyne dressing applications. Data was collected by investigators on Adverse Event Clinical Report Forms for each participant. After initial 12 weeks of application visits, data was collected at 6 month and 12 month (optional) intervals.
Arm/Group | Treated Side | Control Side
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 4/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treated Side (N=12) | Control Side (N=12)
Redness (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Incision Opened (Surgical and medical procedures) | 1 (1) | 0 (0)
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Peeling (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Headaches (General disorders) | 1 (1) | 1 (1)

LIMITATIONS AND CAVEATS:
The Neodyne Dressing is referred to as the "embrace device."

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No